CLINICAL TRIAL: NCT06075888
Title: Evaluation of the Diagnostic Performance of the DISQVER® Metagenomic Sequencing Tool for the Identification of Pathogens in Febrile Neutropenic Haemato-oncology Patients
Brief Title: Metagenomic Sequencing for the Identification of Pathogens in Febrile Neutropenic Patients
Acronym: ADNEMIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: Noscendo (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: ADNEMIA
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Immunodepressed Patients (Hemato-oncology)
Keywords: Neutropenia; Fever; Bacteremia; Viremia; Fungemia; Antibiotic
MeSH Terms: conditions — Neutropenia; Fever; Bacteremia; Viremia; Fungemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Metagenomic diagnosis (mNGS, DISQVER) — Blood sample taken for metagenomic sequencing at inclusion visit.

SUMMARY:
The development of targeted therapies and intensive protocols in oncohaematology has improved the survival of patients with haematological malignancies. The increase in the number of patients treated and their life expectancy has been accompanied by an increase in the incidence of infectious complications secondary to the immunosuppression induced by these therapies.

Febrile neutropenia (NF) is a complication that occurs in approximately 10% to 15% of patients treated for solid tumours and up to 100% of patients treated for haematological malignancies, particularly after bone marrow and/or haematopoietic stem cell transplantation.

In 25% to 30% of cases, NF leads to serious complications. The vast majority of NF cases are caused by microbial infections (bacteria, viruses, fungi, parasites, etc.), which can progress to severe sepsis or septic shock if appropriate treatment is not initiated rapidly (introduction of anti-infective molecules and implementation of associated procedures). If no pathogen is identified during the management of the most severe patients, the prognosis is poor, with a mortality rate of 10%.

The performance of diagnostic strategies is therefore an important factor in improving the prognosis of these patients. To date, the reference diagnosis of microorganisms is based on blood cultures, blood Polymerase Chain Reaction (PCR), β-D-glucan and aspergillosis serology. Identifying the pathogens responsible for NF from a blood sample without an a priori hypothesis and in an optimised timeframe could allow earlier treatment of high-risk NF with implications for management (possible modification of antimicrobial and/or immunosuppressive treatment).

The aim of this study is to evaluate the performance of the mNGS-DISQVER® tool in diagnosing pathogenic microorganisms from blood samples collected from patients being managed for high-risk NF.

DETAILED DESCRIPTION:
1. Clinical context

   The development of targeted therapies and intensive protocols in oncohaematology has improved the survival of patients with haematological malignancies. The increase in the number of patients treated and their life expectancy has been accompanied by an increased incidence of infectious complications secondary to the immunosuppression induced by these therapies.

   Chemotherapy-induced febrile neutropenia (NF) is a common and serious complication occurring in approximately 10% to 15% of patients treated for solid tumours and up to 100% of patients treated for haematological malignancies, particularly after bone marrow transplantation. Febrile neutropenia is defined as a combination of :
   * Neutropenia: neutrophil count <500 g/L or <1000 g/L (if <500 g/L is expected within 48 hours)
   * Fever: >38.5°C on a single occasion or >38°C for more than one hour. NF is associated with high morbidity and mortality (25-30% of serious complications and 10% of mortality). Its occurrence includes the need for hospitalisation with broad-spectrum antibiotic therapy, delayed chemotherapy and loss of opportunity for the patient. In the USA, an episode of NF requiring hospitalisation is associated with an estimated health economic impact of $19,110. A recent study in France estimated the clinical and economic impact of hospitalisation for NF, in terms of number of patients hospitalised, number of stays, in-hospital mortality and average cost per stay, to be €5,333 for haemopathies.

   A significant proportion of NF cases are caused by microbial infections that can progress to septicaemia if probabilistic broad-spectrum antibiotic therapy is not administered within an hour. Furthermore, microbiological documentation remains essential to optimise antibiotic therapy, with blood culture as the reference test. However, this test is limited for a number of reasons: difficulties or slowness in culture, antibiotic treatment prior to sampling, or insufficient sample quantity. Despite the recommended minimum of 3 or 4 pairs of blood cultures, 70% of cases of febrile neutropenia are not microbiologically documented, making it impossible to adapt probabilistic broad-spectrum antibiotic therapy. Another limitation is the time required to obtain results: 6 to 24 hours are required to obtain a positive blood culture, plus another 18 to 24 hours for bacteria to grow on solid media, and another 18 to 24 hours for susceptibility testing (antibiotic susceptibility testing).

   The absence of an identified pathogen in the management of the most severe patients is associated with a poor prognosis, with a mortality rate of 10%. As a result, the performance and timeliness of diagnostic strategies are important factors in improving the prognosis of these patients. In this context, the development of high-throughput sequencing technologies has led to the development of new diagnostic approaches based on the detection of circulating DNA (lcDNA, e.g. used in antenatal screening for trisomy 21). Although more recently democratised, the concept of microbial cDNA is well established in the field of infectious diseases. This technology, based on a blood sample obtained by simple venipuncture, could offer patients with febrile neutropenia an improved diagnosis, particularly in the case of negative blood cultures, and an adjustment in their management.
2. Identification and description of the IVDD

The DISQVERⓇ device is CE-IVD marked according to the In Vitro Diagnostic Directive (IVDD) classification approved until May 2026. The assessment file for its marking according to In-Vitro Diagnostic Regulation (IVDR) is in progress.

DISQVER® is a digital analytical solution developed by Noscendo for the rapid identification of microorganisms in a patient's blood sample from free circulating DNA, without any a priori hypothesis.

The test is based on metagenomic Next Generation Sequencing "mNGS" to identify, without a priori assumptions, the genomic sequences of micro-organisms (bacteria, DNA viruses, fungi and parasites) potentially present in the patient's plasma sample. The genomic sequences identified are then compared with Noscendo's proprietary database of over 16,000 microbial genome sequences, including 1,500 pathogens.

A report detailing all relevant pathogens detected in the sample is provided within a few hours (access to a pseudonymised pdf report according to the laboratory's guidelines, including the micro-organisms found in the highest concentration and the most likely pathogen present).

ELIGIBILITY:
Inclusion Criteria:

* Patient
* Age ≥18 years
* Being treated for solid tumour or haematological malignancy
* Presenting with high-risk febrile neutropenia (high-risk is defined by a Multinational Association for Supportive Care in Cancer (MASCC) score ≥ 21) with an expected duration of neutropenia ≥ 7 days. Neutropenia is defined as an absolute neutrophil count ≤ 500/mm3. Fever is defined as temperature ≥ 38.3°C or ≥ 38°C twice within 1 hour.
* Free, without guardianship, tutelage or subordination;
* covered by a social security scheme or by a third party;
* have given informed consent to participate in the study.

Exclusion Criteria:

* Antibiotic therapy in the 24 hours prior to enrolment, with the exception of prophylactic use of trimethoprim-sulfamethoxazole (Cotrimoxazole) and penicillin G (Oracillin®).
* Previous study participation
* Patients with enhanced protection, i.e. minors, persons deprived of their liberty by a judicial or administrative decision, persons in a health or social care institution, adults under legal protection;
* Pregnant or lactating women of childbearing age (menopause must be documented) who refuse or do not have an effective method of contraception (hormonal/mechanical: per os, injectable, transcutaneous, implantable, intrauterine device or surgical: tubal ligation, hysterectomy, total oophorectomy) for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-01-12 (Estimated); Study Completion 2025-01-12 (Estimated)

PRIMARY OUTCOMES:
Performances (intrinsic diagnostic capabilities) of Metagenomic testing | 1 day
  Based on the microorganisms identified by the conventional work-up and the mNGS-DISQVER® tool, an adjudication committee consisting of a microbiologist, an infectiologist and a haematologist, independent of the study, will assess the presence of at least one pathogen requiring appropriate management. The interpretation of the conventional work-up and that provided by the mNGS-DISQVER® tool will be blinded.
  The intrinsic diagnostic capabilities will be assessed by the sensitivity/specificity of the new mNGS-DISQVER® test, with the classification resulting from the conventional work-up as the reference.

SECONDARY OUTCOMES:
Performances (extrinsic diagnostic capabilities) of Metagenomic testing | 1 day
  The Youden index, the positive and negative predictive values of the new mNGS-DISQVER® test (with conventional work-up as reference) and the proportions of concordant and discordant pairs between the new test and conventional work-up.
Clinical impact of Metagenomic testing on therapeutic choices | 1 day
  The differences between the percentages of patient management modalities (escalation, maintenance, de-escalation or discontinuation of anti-infective treatment) using the mNGS-DISQVER® tool versus the conventional work-up.
Use of Metagenomic testing during clinical patient's management | 1 day
  The mean time taken for conventional assessment, the prevalence of microorganisms diagnosed in routine care (independent of the adjudication committee) and the percentage distribution of anti-infective adjustments according to microorganisms diagnosed in routine care.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - C.H.U. d'Angers, Angers
  - CHU de Brest, Brest
  - C.H.U. de Limoges, Limoges
  - C.H.U. de Poitiers, Poitiers
  - C.H.U. de Tours, Tours

REFERENCES:
- [Derived] Pichon M, Burucoa C; ADNEMIA Study Group. Diagnostic performance of the DISQVER metagenomic sequencing tool for the identification of pathogens in febrile neutropenic patients: the ADNEMIA trial. BMJ Open. 2025 Jan 22;15(1):e087773. doi: 10.1136/bmjopen-2024-087773. PMID 39843376